CLINICAL TRIAL: NCT00074295
Title: Phase II Trial of CG8123, an Autologous Cancer Vaccine (GVAX), in Patients With Selected Stage IIIB and IV Bronchioloalveolar Carcinoma (BAC)
Brief Title: S0310: Vaccine Therapy in Treating Patients With Stage IIIB or Stage IV Bronchoalveolar Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: closed due to lack of availability of vaccine
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000343797; U10CA032102 (NIH); S0310 (Other: SWOG)
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: bronchoalveolar cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): GVAX lung cancer vaccine
  Interventions: Biological: GVAX lung cancer vaccine

INTERVENTIONS:
Biological: GVAX lung cancer vaccine — 6-7 injections per week in rotating locations for five weeks
  Other Names: CG8123

SUMMARY:
RATIONALE: Vaccines made from a person's tumor tissue may make the body build an immune response to kill tumor cells.

PURPOSE: This phase II trial is studying vaccine therapy to see how well it works in treating patients with stage IIIB or stage IV bronchoalveolar (lung) cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression-free and overall survival of patients with selected stage IIIB or stage IV bronchoalveolar carcinoma treated with GVAX lung cancer vaccine.
* Determine the response rate (confirmed and unconfirmed and complete and partial) in patients treated with this vaccine.
* Determine the frequency and severity of toxic effects of this vaccine in these patients.
* Determine the functional status of patients treated with this vaccine.
* Correlate systemic biologic activity (i.e., antigen-specific antitumor and systemic cytokine responses) with clinical outcome in patients treated with this vaccine.

OUTLINE: This is a multicenter study. Patients are stratified according to prior systemic cancer therapy for bronchoalveolar carcinoma (BAC) (yes vs no) and pattern of BAC (diffuse vs nodular).

After successful vaccine manufacturing from tumor tissue procured, patients receive GVAX lung cancer vaccine intradermally (ID) (6-7 injections per vaccination) on weeks 1, 3, 5, 7, and 9 for a total of 5 vaccinations. Treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and at weeks 9, 13, and 21.

Patients are followed at 4 weeks, every 8 weeks for 1 year, and then every 12 weeks for 2 years.

PROJECTED ACCRUAL: A total of 117 patients (67 previously untreated and 50 previously treated) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis* of 1 of the following by radiological features and clinical presentation:

  * Bronchoalveolar carcinoma (BAC)

    * Diffuse or ground glass appearance
  * Adenocarcinoma with bronchoalveolar features
  * BAC with focal invasion NOTE: *Histological confirmation (excluding fine needle aspiration or bronchial brushings or washings) is required after the tumor tissue has been procured and the vaccine has been produced
* Selected stage IIIB (due to malignant pleural effusion) OR stage IV disease
* Measurable or nonmeasurable disease (e.g., diffuse infiltrative process) by CT scan of the chest both before and after tumor tissue procurement for vaccine
* Not a candidate for curative resection
* Tumor accessible for tissue procurement via thoracentesis or a surgical procedure

  * If a pleural effusion is the source of tumor tissue, at least 600 mL of fluid must be available for vaccine manufacture
  * Resection of brain metastases may be used for vaccine processing

    * Surgery must be done after study entry
* Asymptomatic previously treated (e.g., surgical resection or radiotherapy) brain metastases allowed provided the patient is neurologically stable
* No active or impending spinal cord compression or evidence of pericardial tamponade

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* CD4 count greater than 200/mm^3
* No bleeding disorder

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN) (3 times ULN if liver metastases are present)
* SGOT or SGPT no greater than 2.5 times ULN (5 times ULN if liver metastases are present)
* Alkaline phosphatase no greater than 2.5 times ULN (5 times ULN if bone metastases are present)

Renal

* Not specified

Cardiovascular

* See Disease Characteristics
* Patients requiring surgery for tumor tissue procurement must meet the following criteria:

  * Pulmonary artery systolic pressure < 40 mm Hg by echocardiogram*
  * LVEF > 40%
* No symptomatic congestive heart failure
* No thrombolic disorder
* No unstable angina pectoris
* No cardiac arrhythmia NOTE: *Not needed if patient has no tricuspid regurgitation

Pulmonary

* No pulmonary hypertension
* No significant baseline hypoxia (i.e., O_2 saturation less than 90% OR requires greater than 2 L/min of supplemental O_2 via nasal cannula) by an oxygen saturation test
* No postobstructive pneumonia
* Patients requiring thoracoscopic surgery or thoracotomy for tumor tissue procurement must meet the following criteria:

  * Alveolar partial pressure of CO_2 < 45 mm Hg
  * Predicted postresection FEV_1 ≥ 1.0 L
  * DLCO > 50% of predicted

Immunologic

* No active immune or autoimmune disease
* No systemic lupus erythematosus
* No sarcoiditis
* No rheumatoid arthritis
* No glomerulonephritis
* No vasculitis
* No serious infection
* No hypersensitivity to any of the following:

  * Sargramostim (GM-CSF)
  * Pentastarch
  * Gentamicin
  * Human serum albumin
  * Dimethyl sulfoxide
  * Porcine trypsin
  * Fetal bovine serum
  * Recombinant benzonase
  * Other components of the vaccine or CG6444 adenoviral vector used in this study

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No poor nutritional status
* No psychiatric illness or social situation that would preclude study compliance or increase operative risk
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission
* No other concurrent uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior biologic therapy
* No prior gene therapy, including adenoviral-based therapy

Chemotherapy

* More than 4 weeks since prior chemotherapy

  * No prior regional chemotherapy administered through the pulmonary artery (if resection of the tumor in the treated lobe is planned)

Endocrine therapy

* More than 14 days since prior systemic corticosteroids
* No concurrent steroids

Radiotherapy

* See Disease Characteistics
* More than 4 weeks since prior radiotherapy

  * Disease must be outside the areas of prior radiotherapy OR clear progression at prior irradiated sites must be documented
* No prior radiotherapy to the tumor mass targeted for resection

Surgery

* See Disease Characteristics
* More than 7 days since prior surgery and recovered

Other

* More than 2 weeks since prior epidermal growth factor receptor inhibitors
* No other concurrent nonprotocol-specified treatment
* No concurrent immunosuppressants
* No concurrent chronic anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Progression-free and overall survival
Response rate
Toxicity
Functional status
Correlation of systemic biologic activity with clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Angela Davies, MD, Principal Investigator — University of California, Davis; Raja Mudad, MD, FACP, Principal Investigator — Tulane University Health Sciences Center